CLINICAL TRIAL: NCT03054805
Title: The Effect of Probiotics on Constipation, and Intestinal Microflora in Children With Functional Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103-0519A3
Record Dates: First submitted 2017-01-17; First posted 2017-02-16 (Actual); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2014-09

CONDITIONS: Functional Constipation
MeSH Terms: interventions — Magnesium Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Magnesium oxide and MIYAIRI-BM (Experimental): Magnesium oxide 125 mg twice per day for children with weight < 15 kg, 250 mg twice per day for weight <15-30 kg, and 500 mg twice per day for weight > 30 kg for 12 weeks.
  MIYAIRI-BM 1 package (1g) divided as 0.5 g twice per day for children with weight < 15 kg, 2 packages divided as 1 g twice per day for weight 15-30 kg, and 3 packages divided as 1.5 g twice per day for weight > 30 kg for 12 weeks.
  Interventions: Drug: Magnesium Oxide; Drug: MIYAIRI-BM
- Magnesium oxide (Active Comparator): MIYAIRI-BM 1 package (1g) divided as 0.5 g twice per day for children with weight < 15 kg, 2 packages divided as 1 g twice per day for weight 15-30 kg, and 3 packages divided as 1.5 g twice per day for weight > 30 kg for 12 weeks.
  Interventions: Drug: Magnesium Oxide
- Healthy Children (No Intervention): Healthy Children

INTERVENTIONS:
Drug: Magnesium Oxide — Magnesium oxide 250 mg per day for children with weight < 15 kg, 500 mg per day for weight <15-30 kg, and 1000 mg per day for weight > 30 kg
  Other Names: MgO
  Arms: Magnesium oxide; Magnesium oxide and MIYAIRI-BM
Drug: MIYAIRI-BM — MIYAIRI-BM 1 g (1package) per day for children with weight < 15 kg, 2g per day for weight 15-30 kg, and 3g per day for weight > 30 kg
  Other Names: Clostridium Butyricum MIYAIRI
  Arms: Magnesium oxide and MIYAIRI-BM

SUMMARY:
To compare the differences of fecal microflora between constipated and non-constipated healthy children, and evaluate the efficacy of probiotics in reducing symptoms of constipation and the influence of intestinal microflora in children with functional constipation.

DETAILED DESCRIPTION:
The investigators performed a monocentric, prospective, randomized controlled trial including 120 pediatric patients (aged 6 months - 10 years old) with functional constipation and 30 healthy age-matched healthy children as control. The investigators shall evaluate the children according to the Rome III Diagnostic Criteria for functional constipation.

The 120 enrolled patients are randomized in to two groups: Group A receiving magnesium oxide and probiotics (MIYAIRI-BM), Group B receiving only magnesium oxide. Each patient is assigned the evaluation constipation symptoms and detection of microflora (beneficial and harmful bacteria) in fecal samples at the enrollment, 4 weeks, and 12 weeks. Patients who take less than 80% of the appropriate dose of medications are withdrawn from the study. All patients included in the study will be given informed oral consent before entering the study.

The data of the fecal microflora evaluated in 60 healthy children are used as control.

ELIGIBILITY:
Inclusion Criteria:

Rome III Diagnostic Criteria for functional constipation for children aged 6 months - 4 years old is as the following:

1. Two or fewer defecations per week.
2. At least one episode per week of incontinence after acquiring toileting skills.
3. History of excessive stool retention.
4. History of painful or hard bowel movements.
5. Presence of a large fecal mass in the rectum.
6. History of large-diameter stools that may obstruct the toilet. Children aged 6 months - 4 years old is evaluated as functional constipation if two of the situations mentioned above lasted for one month.

Rome III Diagnostic Criteria for functional constipation for children aged 4 years old and above is as the following:

1. Two or fewer defecations in the toilet per week.
2. At least one episode of fecal incontinence per week.
3. History of retentive posturing or excessive volitional stool retention.
4. History of painful or hard bowel movements.
5. Presence of a large fecal mass in the rectum.
6. History of large diameter stools that may obstruct the toilet. Children aged 4 years old and above is evaluated as functional constipation if two of the situations mentioned above happens at least once per week

Exclusion Criteria:

1. gastroesophageal reflux disease
2. inflammatory bowel disease
3. cardiopulmonary diseases
4. liver disease
5. renal disease
6. genetic diseases
7. endocrinal diseases
8. received abdominal surgeries

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2016-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial is expected to recruit 180 children, but the actual willingness to participate in the trial is 153 children.
Groups:
- Magnesium Oxide and MIYAIRI-BM: Magnesium oxide 125 mg twice per day for children with weight < 15 kg, 250 mg twice per day for weight <15-30 kg, and 500 mg twice per day for weight > 30 kg for 12 weeks.
  MIYAIRI-BM 1 package (1g) divided as 0.5 g twice per day for children with weight < 15 kg, 2 packages divided as 1 g twice per day for weight 15-30 kg, and 3 packages divided as 1.5 g twice per day for weight > 30 kg for 12 weeks.
  Magnesium Oxide: Magnesium oxide 250 mg per day for children with weight < 15 kg, 500 mg per day for weight <15-30 kg, and 1000 mg per day for weight > 30 kg
  MIYAIRI-BM: MIYAIRI-BM 1 g (1package) per day for children with weight < 15 kg, 2g per day for weight 15-30 kg, and 3g per day for weight > 30 kg
- Healthy Children: Healthy children without any treatment
Period: Overall Study
Arm/Group | Magnesium Oxide and MIYAIRI-BM | Magnesium Oxide | Healthy Children
Started | 58 | 51 | 44
Completed | 42 | 41 | 42
Not Completed | 16 | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Oxide and MIYAIRI-BM | Magnesium Oxide | Healthy Children | Total
Number analyzed (Participants) | 42 | 41 | 42 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 41 | 42 | 125
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.75 (1.25) | 3.92 (1.83) | 4.08 (2.41) | 3.58 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 17 | 64
  Male | 18 | 18 | 25 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change of Clostridium Butyricum Miyairi Expression After Probiotics Supplementation in Constipated Children.
Description: The expression of Clostridium butyricum Miyairi (CBM) in constipated children feces means a better outcome measure.
Time Frame: Change from baseline Clostridium butyricum Miyairi expression at 3 months.
Measure: Mean (Standard Deviation); unit: number of bacteria per mg of feces
Arm/Group | Magnesium Oxide and MIYAIRI-BM | Magnesium Oxide | Healthy Children
Number analyzed (Participants) | 42 | 41 | 42
number of bacteria per mg of feces | 0.00486 (0.00696) | 0.0000148 (0.0000266) | 0.00000189 (0.00000341)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Magnesium Oxide and MIYAIRI-BM | Magnesium Oxide | Healthy Children
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/51 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/51 | 0/44
Other Adverse Events (participants affected / at risk) | 0/58 | 0/51 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No